CLINICAL TRIAL: NCT03627247
Title: Impact of a Cognitive Behavioral Stress Management Intervention on Cortisol Regulation During Pregnancy
Brief Title: Impact of Stress Management on Cortisol Patterns in Low-Income Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Guido Urizar, Professor, California State University, Long Beach
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07373610
Record Dates: First submitted 2018-07-27; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy Related; Stress, Physiological
Keywords: cognitive behavioral; stress management; pregnancy; cortisol

STUDY DESIGN:
Intervention Model Description: prospective, pre-test post-test, experimental control group design
Who Masked: Outcomes Assessor
Masking Description: Staff completing assessments were blind to participants' study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Stress Management (Experimental): Women randomized to CBSM participated in an eight-week prenatal course called SMART Moms (Stress Management and Relaxation Training for Moms) aimed at teaching coping and relaxation skills that address stressors and daily challenges experienced during pregnancy and motherhood.
  Interventions: Behavioral: Cognitive Behavioral Stress Management
- Attention Control Group (No Intervention): Women randomized to the AC group participated in an eight-week program where they received printed materials (offered in Spanish and English) by mail once per week, on common prenatal health information topics (e.g., common discomforts of pregnancy, labor and delivery) chosen from the March of Dimes Foundation's "Becoming a Mom" handouts (March of Dimes, 2011). Women in this group were contacted once per week by phone by a research staff member to make sure that they received their mailed prenatal health information and to see if they had any questions.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management — Interactive activities (e.g., role-playing, use of physical props to introduce concepts related to coping and stress) were designed for each class to optimize participant engagement and understanding of the course material while tailoring class content to the stressors commonly reported by participants. Each week, participants were given coping and relaxation skills to practice at home (e.g., cognitive reappraisal, diaphragmatic breathing) and were asked to record their experiences on an activity log that was collected and discussed in class the following week. Course content was taught from a detailed training manual (Urizar & Kofman, 2012).
  Arms: Cognitive Behavioral Stress Management

SUMMARY:
PROJECT NARRATIVE: As demonstrated by a growing number of studies, experiencing high levels of stress during pregnancy, including elevated levels of the stress hormone cortisol, can lead to significant long-term health problems for mothers and their infants. The objective of the proposed research is to test whether an innovative stress management intervention, offered during pregnancy, is effective in reducing stress and cortisol levels among low-income pregnant women. The results of the proposed work have substantial public health implications in helping to prevent the onset of stress-related health complications among mothers and their infants.

DETAILED DESCRIPTION:
PROJECT SUMMARY: As demonstrated by a growing number of studies, stress experienced during pregnancy can lead to significant long-term health problems for mothers and their infants. One biological mechanism that has been identified in heightening a woman's risk for developing stress-related health complications during pregnancy and the postpartum period is the stress hormone cortisol. However, the best methods for regulating cortisol, in order to optimize maternal and infant health outcomes, have received little attention. The objective of the proposed research is to conduct a two-arm, pilot randomized controlled study to test the efficacy of a prenatal cognitive behavioral stress management (CBSM) intervention in regulating cortisol and stress levels among low-income pregnant women. A total of 100 women will be randomized to either a group-based, 8-week prenatal CBSM arm (i.e., cognitive coping and relaxation skills training) or a standard-of-care comparison arm (i.e., usual pre- and postnatal care) to examine whether women receiving the CBSM intervention will have significantly lower cortisol output and stress levels, relative to women randomized to the standard-of-care comparison arm. This study will also examine whether these decreases in cortisol and stress levels are mediated through behavior change processes (e.g., increased self-efficacy and use of cognitive coping and relaxation skills). This hypothesis has been formulated on the basis of preliminary data collected by the principal investigator and study collaborators. Through formative research, this pilot work will develop and empirically test a prenatal CBSM stress management intervention among low-income pregnant women for use in local prenatal centers. The results of the proposed work have substantial public health implications and are expected to advance the investigator's understanding of how pregnant women effectively use these cognitive coping and relaxation skills to adopt healthy behaviors and produce change that can positively impact their health, as well as that of their infant. Further, the proposed research will yield a CBSM intervention that can be readily delivered in community settings, is scalable, and is relatively low cost. Finally, these results will help identify those subgroups of pregnant women that may do particularly well (or poorly) with these innovative approaches to stress management. This has important implications for the tailoring of CBSM programs to individual needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* less than 17 weeks pregnant
* fluent in either Spanish or English

Exclusion Criteria:

* Major medical problems (e.g., gestational diabetes, major depression)
* Taking medications that may interfere with cortisol levels (e.g., asthma inhaler, antidepressants).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2014-08-30 (Actual); Study Completion 2014-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Overall Salivary Cortisol Output during Pregnancy and Early Postpartum calculated from seven saliva samples collected on one collection day at each study time point. | Salivary cortisol assessments were conducted at baseline, during the second trimester (i.e., upon completing the eight-week program), third trimester (between 30-32 weeks of pregnancy), and at three months post partum.
  The overall amount of cortisol secreted throughout the day was computed using area under the curve (AUC) in nmol/L. Larger numbers of AUC represent a greater amount of cortisol produced throughout the day. Elevated overall cortisol secretion throughout the day (AUC) has been associated with a number of adverse health outcomes. Change in AUC will be examined using mixed methods models throughout each study time point.
Change in Cortisol Awakening Response during Pregnancy and Early Postpartum calculated from seven saliva samples collected on one collection day at each study time point. | Salivary cortisol assessments were conducted at baseline, during the second trimester (i.e., upon completing the eight-week program), third trimester (between 30-32 weeks of pregnancy), and at three months post partum.
  The cortisol awakening response (CAR) was computed using the percent increase in morning cortisol in nmol/L. CAR measures the acute rise in cortisol typically seen after waking in the morning with larger numbers representing a greater percent increase in cortisol from waking to 30 minutes after waking. An altered CAR has been associated with a number of adverse health outcomes. Change in CAR will be examined used mixed methods models throughout each study time point.
Change in Diurnal Cortisol Slope during Pregnancy and Early Postpartum calculated from seven saliva samples collected on one collection day at each study time point. | Salivary cortisol assessments were conducted at baseline, during the second trimester (i.e., upon completing the eight-week program), third trimester (between 30-32 weeks of pregnancy), and at three months post partum.
  Diurnal cortisol slope was estimated by calculating the change in cortisol from waking to 8PM in nmol/L, with larger numbers representing a flatter diurnal cortisol slope (i.e., smaller decrease in cortisol levels across the day). A flatter diurnal cortisol slope has been associated with a number of adverse health outcomes. Change in diurnal cortisol slope will be examined using mixed methods models throughout each study time point.

SECONDARY OUTCOMES:
Change in Perceived Stress during Pregnancy and Early Postpartum. One total perceived stress score will be calculated using Cohen's Perceived Stress Scale, which is a questionnaire completed by participants at each study time point. | Perceived stress assessments were conducted at baseline, during the second trimester (i.e., upon completing the eight-week program), third trimester (between 30-32 weeks of pregnancy), and at three months post partum.
  Perceived stress was assessed using the 14-item version of the Perceived Stress Scale (PSS-14; Cohen & Williamson, 1988). The PSS-14 measures the degree to which situations in one's life over the past month were appraised as stressful, with higher scores (range = 0-56) reflecting higher stress levels. The PSS-14 has shown good test-retest reliability and internal consistency in both general and pregnancy populations (Huizink et al., 2002) and has demonstrated sensitivity to changes in the perceived stress levels of pregnant women receiving a relaxation intervention (Bastani et al., 2005). The PSS-14 demonstrated good internal consistency across the four time points in the current study (α range = 0.74-0.75). Change in total perceived stress will be examined used mixed methods models throughout each study time point.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Urizar, PhD, Principal Investigator — California State University, Long Beach

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the questions asked in this study, survey respondents were assured raw data would remain confidential and would not be shared.
  Data not available / The data that has been used is confidential

REFERENCES:
- [Result] Scheyer K, Urizar GG Jr. Altered stress patterns and increased risk for postpartum depression among low-income pregnant women. Arch Womens Ment Health. 2016 Apr;19(2):317-28. doi: 10.1007/s00737-015-0563-7. Epub 2015 Aug 15. PMID 26275372